CLINICAL TRIAL: NCT02202941
Title: Effect of Procalcitonin-guided Treatment on Duration of Antibiotic Therapy and Cost in Septic Patients in Korea
Brief Title: Procalcitonin-guided Treatment on Duration of Antibiotic Therapy and Cost in Septic Patients
Acronym: PRODA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: National Evidence-based healthcare Collaborating Agency (NECA) (Unknown); Asan Medical Center (Other); Samsung Medical Center (Other); Severance Hospital (Other)
Responsible Party: Principal Investigator, Sang-Min Lee, Associate professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRODA-2014
Record Dates: First submitted 2014-07-24; First posted 2014-07-29 (Estimated); Last update posted 2018-11-02 (Actual); Status verified 2018-11

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Procalcitonin guided treatment (Experimental): Patients who will be randomized to this arm will receive antibiotics therapy based on procalcitonin-guided algorithm.
  Interventions: Other: Procalcitonin guided treatment
- Conventional treatment (Active Comparator): Patients who will be randomized to this arm will receive antibiotic therapy based on conventional practice.
  Interventions: Other: Conventional treatment

INTERVENTIONS:
Other: Procalcitonin guided treatment — Patients who will be randomized to arm will receive antibiotics therapy based on procalcitonin measurement on day 1, 3, 5, 7, 9, 11 and 13.
  Arms: Procalcitonin guided treatment
Other: Conventional treatment — Patients who will be randomized to this arm will receive antibiotic therapy based on conventional practice.
  Arms: Conventional treatment

SUMMARY:
This clinical trial is aimed to show a procalcitonin-guided treatment algorithm may shorten duration of antibiotic therapy safely and cost-effectively in sepsis patients of Korean ICU.

ELIGIBILITY:
Inclusion Criteria:

* All patients with suspicious or confirmed sepsis at admission or during stay in ICU
* Patients with antibiotic duration of less than 48 hours before enrollment

Exclusion Criteria:

* Age less than or equal to 18 years
* Known pregnancy
* Specific infections for which long-term antibiotic treatment for 3 weeks more is strongly recommended: infective endocarditis, empyema, osteomyelitis et al.
* severe immunocompromised patients : HIV infected patients (CD4 count < 200 cells/mm3), Neutropenia (ANC count < 500/mm3)
* Presence of do-not-resuscitate order

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2015-02 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Duration of antibiotic treatment | up to 28 days

SECONDARY OUTCOMES:
Clinical response to treatment for infection | up to 28 days
  success vs failure vs relapse after treatment
In ICU mortality | up to 28 days
All cause mortality | up to 28 days
In hospital mortality | up to 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Sang-Min Lee, M.D., Principal Investigator — Seoul National University Hospital
Locations (4):
- South Korea (4):
  - Seoul National University Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Asan Medical Center, Seoul
  - Severance Hospital, Seoul

REFERENCES:
- [Derived] Jeon K, Suh JK, Jang EJ, Cho S, Ryu HG, Na S, Hong SB, Lee HJ, Kim JY, Lee SM. Procalcitonin-Guided Treatment on Duration of Antibiotic Therapy and Cost in Septic Patients (PRODA): a Multi-Center Randomized Controlled Trial. J Korean Med Sci. 2019 Apr 15;34(14):e110. doi: 10.3346/jkms.2019.34.e110. PMID 30977312